CLINICAL TRIAL: NCT04951856
Title: Acute Myocardial Infarction Upbound to PCI Immediately (STEMI) or in the Next Three Days (NSTEMI), and Randomized to Subcutaneous Evolocumab or Normal Strategies to Reach Guidelines LDL Objectives in the Real-world - The AMUNDSEN-real Study
Brief Title: Evolocumab or Normal Strategies to Reach LDL Objectives in Acute Myocardial Infarction Upbound to PCI
Acronym: AMUNDSEN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action Research Group (Other); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP201075; 2021-000573-80 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-07-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI
Keywords: STEMI; NSTEMI; PCI; STATIN; EVOLOCUMAB; Anti-PCSK9; LDL-C
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — evolocumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evolocumab + SOC (Experimental): Investigational Product is open label Evolocumab (Repatha®) 140 mg every two weeks: first subcutaneous injection at the time of randomization, before PCI, followings during 12 months.
  Interventions: Drug: Evolocumab 140 MG/ML
- Standard of care (SOC) (Active Comparator): management as recommended in ESC/EAS 2019 guidelines, within reimbursement criteria
  Interventions: Drug: Standard of care (SOC)

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML — Evolocumab (Repatha®) 140 mg every two weeks: first subcutaneous injection at the time of randomization, before PCI, followings during 12 months.
  Other Names: Repatha
  Arms: Evolocumab + SOC
Drug: Standard of care (SOC) — management as recommended in ESC/EAS 2019 guidelines, within reimbursement criteria
  Arms: Standard of care (SOC)

SUMMARY:
AMUNDSEN-real is a phase IV, international (7 European countries), multicenter, controlled, open label study randomized, in 2 parallel groups of patients with a diagnosis of STEMI or NSTEMI with an indication for PCI, using the PROBE study design (Prospective Randomised Open, Blinded Endpoint).

The objective of this study is to demonstrate the superiority of evolocumab versus standard of care in reaching a LDL-C reduction of ≥ 50% from baseline and a LDL-C goal of <1.4 mmol/L (<55 mg/dL) at 12 months follow-up on the overall population.

Central randomization uses an IWRS. Stratification is by center and stratum with random block size, generated according to the procedures of the sponsor, by a statistician not involved in the study.

DETAILED DESCRIPTION:
Previous randomized studies and several meta-analyses have shown a positive effect of high-dose statins pretreatment on peri-procedural Myocardial Infarction (MI) incidence with favorable trends on mortality in both Acute Coronary Syndrome (ACS) and stable Coronary Artery Disease patients.

Numerous epidemiological studies, Mendelian randomization studies, and Randomized Controled Trials have consistently demonstrated a log-linear relationship between the absolute changes in plasma LDL-C and the risk of Cardio-Vascular (CV) disease. The effect of LDL-C on the risk of a new CV event appears to be determined by the absolute magnitude, the duration of exposure to LDL-C and possibly the time to reach the recommended target of low LDL in ACS patients.

There are good reasons to believe that the Proprotein Convertase Subtilisin/Kexin type 9 (PCSK9) inhibitors could provide additional benefits when used early in MI patients treated with PCI revascularization.

That's why the hypothesis of AMUNDSEN study is to demonstrate the superiority of a strategy using evolocumab before PCI in STEMI or NSTEMI patients versus standard of care (SOC) as described in the 2019 European Society of Cardiology / European Atherosclerosis Society (ESC/EAS) guidelines on dyslipidemia, to reach a Low-Density Lipoprotein Cholesterol (LDL-C) reduction of ≥ 50% from baseline and a LDL-C goal of <1.4 mmol/L (<55 mg/dL) at the end of the study (LDL targets of the 2019 ESC/EAS guidelines).

ELIGIBILITY:
Inclusion Criteria:

Participant meeting all of the following criteria will be considered for enrolment into the trial:

1. Male or female
2. Diagnosis of STEMI or NSTEMI

   STEMI defined as:
   * symptoms of acute MI of at least 30 min AND
   * within the previous 24 hours with new persistent ST-segment elevation ≥1 mm in ≥2 continuous ECG leads AND
   * an indication for primary PCI AND
   * > 55 years reported by the patient

   NSTEMI defined as:
   * Age≥18
   * a history of chest discomfort or ischemic symptoms of ≥10 minutes duration at rest ≤48 hours prior to entry into the trial with no evidence of persistent ST-segment elevation and with an elevated troponin (≥ the upper limit of normal according to local laboratory norms), AND
   * indication for a coronary angiogram within 72hrs AND
   * indication for PCI AND
   * at least one the following high-risk characteristics: Diabetes Peripheral Artery Disease Multivessel (≥ 2 or LM) disease on the coronary angiogram History of MI or stroke without sequels prior to randomization eGFR: 15 to 45 mL/min/1.73 m2 calculated with MDRD formula at randomization
3. Statin at maximal tolerated dose, as part of the standard of care at randomization, means Intent to treat with statin and the patient will receive his first dose as soon as possible after admission
4. Informed consent obtained in writing at enrolment into the trial

Exclusion Criteria:

Participant presenting with any of the following will not be included in the trial:

1. Fibrinolysis treatment
2. Planned CABG
3. Ongoing hemodynamic instability defined as any of the following:

   * Killip Class III or IV
   * Sustained and/or symptomatic hypotension (systolic blood pressure < 80 mm Hg)
   * Known left ventricular ejection fraction < 30%
4. Evidence of severe hepatobiliary disease: current active hepatic dysfunction or active biliary obstruction, decompensated cirrhosis or infectious/inflammatory hepatitis
5. Active malignancy
6. A comorbid condition with an estimated life expectancy of ≤ 12 months
7. Previously received or receiving evolocumab or any other therapy to inhibit PCSK9
8. Known sensitivity to any of the products or components to be administered during trial
9. Female subject is pregnant, had a positive pregnancy test at inclusion, breastfeeding, or planning to become pregnant or breastfeed during treatment and for an additional 17 weeks after the last dose of IMP
10. Currently receiving treatment in any other investigational device or drug trial, or less than 30 days since ending treatment on another investigational device or drug trial.
11. Participant likely to not be available to complete all protocol-required trial visits or procedures, and/or to comply with all required trial procedures to the best of the participant and investigator's knowledge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2166 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2028-05-22 (Estimated)

PRIMARY OUTCOMES:
LDL-C reduction of ≥ 50% from baseline and a final LDL-C of <1.4 mmol/L (<55 mg/dL) at 12 months follow-up. | From baseline and at 12 months
  Monitoring of changes in LDL-C levels

SECONDARY OUTCOMES:
LDL-C reduction of ≥ 50% from baseline and a final LDL-C of <1.4 mmol/L (<55 mg/dL) at 12 months follow-up, country by country. | From baseline and at 12 months
  The same rules as above for the primary endpoint, will apply.
LDL-C reduction of ≥ 50% and an LDL-C goal of <1.4 mmol/L (<55 mg/dL)and other relevant thresholds: <70, <40, and <20 mg/dL | From baseline to 6 weeks and 22 weeks, 12, 24 months and end-of-follow-up(longest follow up for each patient)
  Monitoring of changes in LDL-C levels
Percent change in levels of LDL-C | From baseline to 6 weeks, 22 weeks, 12, 24 months, and end of follow-up(longest follow up for each patient)
  Monitoring of changes in LDL-C levels
Time to achieve LDL-C target | Up to 12 months
  Monitoring of changes in LDL-C levels
Time averaged LDL-C change | Up to 12 months, at 24 months, and end of follow-up(longest follow up for each patient)
  Monitoring of changes in LDL-C levels
Change on total cholesterol | At baseline, 6 weeks, 22 weeks, 12, 24 months, and end of follow-up(longest follow up for each patient)
  Monitoring of changes in cholesterol levels
Change on HDL-C | At baseline, 6 weeks, 22 weeks , 12, 24 months, and end of follow-up(longest follow up for each patient)
  Monitoring of changes in HDL-C levels
Change on triglycerides | At baseline, 6 weeks, 22 weeks, 12, 24 months, and end of follow-up(longest follow up for each patient)
  Monitoring of changes in triglycerides levels
Change on non-HDL-C | At baseline, 6 weeks, 22 weeks, 12, 24 months, and end of follow-up(longest follow up for each patient)
  Monitoring of changes in non-HDL-C levels
Lipoprotein(a) (Lp(a) | at 12 months.
  Monitoring of (Lp(a)

OTHER OUTCOMES:
Composite of death or any hospitalization for a Cardiovascular (CV) reason | from randomization to 12, 24 months, and end of follow-up (longest follow up for each patient)
  Data obtained from reported adverse events occurred during participation to the study
Composite of death, MI, stroke, unplanned revascularization | from randomization to 12, 24 months, and end of follow-up (longest follow up for each patient)
  Data obtained from reported adverse events occurred during participation to the study
Individual endpoints of the composite endpoint above (death, MI, Stroke, unplanned revascularization) | from randomization to 12, 24 months, and end of follow-up (longest follow up for each patient)
  Data obtained from reported adverse events occurred during participation to the study
Pooled analysis of relationship between time to achieve LDL-C goal and death or any hospitalization for a CV reason | from randomization to 12, 24 months, and end of follow-up (longest follow up for each patient)
  Data obtained from reported adverse events occurred during participation to the study and LDL-C levels

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MONTALESCOT, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- ACTION Group, Institut de Cardiologie, Centre Hospitalier Universitaire Pitié Salpêtrière (APHP), UPMC, Paris, France